CLINICAL TRIAL: NCT04309383
Title: Assessment of ShuntCheck Performance Characteristics in Asymptomatic Patients With Pseudotumor Cerebri
Brief Title: ShuntCheck Performance Characteristics in Asymptomatic Pseudotumor Cerebri Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: NeuroDx Development (Industry)
Responsible Party: Principal Investigator, Naomi Abel, Assistant Professor, College of Medicine Neurosurgery, University of South Florida
Other Study IDs: Pro00042422
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pseudotumor Cerebri
Keywords: Pseudotumor Cerebri, Ventriculoperitoneal Shunt
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ShuntCheck: Participants will be administered the ShuntCheck diagnostic test.
  Interventions: Diagnostic Test: ShuntCheck

INTERVENTIONS:
Diagnostic Test: ShuntCheck — The intervention is an FDA-cleared device utilizing a transcutaneous thermal convection to analyze shunt flow.

SUMMARY:
The purpose of the study is to determine if the ShuntCheck test can correctly identify flow or no flow in a ventriculoperitoneal shunt in patients with pseudotumor cerebri.

DETAILED DESCRIPTION:
The purpose of the study is to determine if the ShuntCheck test can correctly identify flow or no flow in a ventriculoperitoneal shunt in patients with pseudotumor cerebri.

Flow may be limited due to slit ventricles

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older Adult men or women who possess a VP shunt placed for PTC;
* Capable of providing valid signed informed consent, or has a legal guardian, health care agent, or surrogate decision maker (according to local statutes, and collectively referred to as "surrogates" in this protocol) capable of providing valid, signed informed consent;
* Subjects will be asymptomatic visiting for routine care at 2-4 weeks post op

Exclusion Criteria:

* Presence of multiple shunts, or presence of more than one distal shunt catheter (regardless of function) crossing the clavicle ipsilateral to the shunt with suspected obstruction;
* ShuntCheck test would interfere with standard patient care, or emergency shunt surgery that cannot be delayed is indicated;
* Presence of an interfering open wound or edema over any portion of the VP shunt.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of asymptomatic PTC research subjects who have a VP shunt with a single ventricular catheter implanted for PTC and are visiting for routine care.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-10-29 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Specificity of ShuntCheck test | 15 minutes
Negative Predictive Value of ShuntCheck test | 15 minutes

SECONDARY OUTCOMES:
Specificity of performing ShuntCheck test twice | 60 minutes
Negative Predictive Value of performing ShuntCheck test twice | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Abel, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida Department of Neurological Surgery and Brain Repair, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
At present there is no plan to share any individual participant data.